CLINICAL TRIAL: NCT06338059
Title: Relationship Between Vitamin D and Vitamin B12 Levels and Neuropathic Pain in Lipedema:Cross Sectional Study
Brief Title: Relationship Between Vitamin D and Vitamin B12 Levels and Neuropathic Pain in Lipedema
Status: Active, not recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Gulcanozturkchatipchousein
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Vitamin D Deficiency; B12 Deficiency Vitamin; Lipedema
Keywords: Vitamin D, B12 Deficiency Vitamin,Lipedema,Pain
MeSH Terms: conditions — Vitamin D Deficiency; Vitamin B 12 Deficiency; Lipedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- painDETECT questionnaire scores> 13 likely or possible neuropathic pain (group 1): lipedema patients showing NP symptoms
  Interventions: Other: Vitamin B12 Level
- painDETECT questionnaire scores13 unlikely neuropathic pain(group 2): lipedema patients showing no NP symptoms
  Interventions: Other: Vitamin B12 Level

INTERVENTIONS:
Other: Vitamin B12 Level — Vitamin B12 Level Laboratory measurement of patient's vitamin B12 level in unit of pg/mL 25 OH Vitamin D Level Laboratory measurement of patient's 25 OH vitamin D level in unit of ng/dl
  Other Names: 25 OH Vitamin D Level

SUMMARY:
Lipedema is a disease characterized by bilateral abnormal fat deposition in the upper and lower extremities. Pain is a common symptom in lipedema.Vitamin D plays an important role in chronic pain. Vitamin B have analgesic role in some neuropathic pain conditions.This study aimedto evaluate the relationship between vitamin D and vitamin B12 levels and neuropathic pain in lipedema.

DETAILED DESCRIPTION:
In this cross sectional study 200 lipedema patients will beincluded. According to painDETECT questionnaire scores of cases with lipedema patients will be divided into two groups;An overall score of > 13 likely or possible neuropathic pain (group 1) and <13 unlikely NP (group 2). Patients' age, gender, comorbid diseases and laboratory values (25 OH vitamin D and vitamin B12 levels) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* The patients diagnosed byan experienced physical medicine and rehabilitation specialist for the diagnosis of lipedema

Exclusion Criteria:

* individuals who did not have 25(OH)D and B12 values in the past 6 months,
* those with a history of gastrectomy or bypass surgery,
* those consuming a vegetarian diet, those with lymphedema or chronic venous insufficiency, endocrine diseases, rheumatic diseases, malignancy, neurological diseases, and musculoskeletaldiseases that can be related to lower extremity neuropathic or nociceptivepain.

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: lipedema patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin B12 Level | 1 day
  Laboratory measurement of patient's vitamin B12 level in unit of pg/mL
25 OH Vitamin D Level | 1 day
  Laboratory measurement of patient's 25 OH vitamin D level in unit of ng/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Gulcan Ozturk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Poojari A, Dev K, Rabiee A. Lipedema: Insights into Morphology, Pathophysiology, and Challenges. Biomedicines. 2022 Nov 30;10(12):3081. doi: 10.3390/biomedicines10123081. PMID 36551837
- [Result] Kiraly SJ, Kiraly MA, Hawe RD, Makhani N. Vitamin D as a neuroactive substance: review. ScientificWorldJournal. 2006 Jan 26;6:125-39. doi: 10.1100/tsw.2006.25. PMID 16493517
- [Result] Gharibpoor F, Ghavidel-Parsa B, Sattari N, Bidari A, Nejatifar F, Montazeri A. Effect of vitamin B12 on the symptom severity and psychological profile of fibromyalgia patients; a prospective pre-post study. BMC Rheumatol. 2022 Sep 1;6(1):51. doi: 10.1186/s41927-022-00282-y. PMID 36045399